CLINICAL TRIAL: NCT02586987
Title: A Phase I, Open-Label, Multi-Centre Study to Assess the Safety, Tolerability and Preliminary Anti-tumour Activity of Ascending Doses of Selumetinib (AZD6244 Hyd-sulfate) in Combination With MEDI4736 and Selumetinib in Combination With MEDI4736 and Tremelimumab in Patients With Advanced Solid Tumours
Brief Title: A Study to Assess the Safety, Tolerability and Anti-tumour Activity of Ascending Doses of Selumetinib in Combination With MEDI4736 and Selumetinib in Combination With MEDI4736 and Tremelimumab in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1345C00003
Record Dates: First submitted 2015-09-21; First posted 2015-10-27 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Lung Cancer; Melanoma; Head and Neck Carcinoma; Gastroesophageal Cancer; Breast Cancer; Pancreatic Adenocarcinoma; Colorectal Cancer; Biliary Tract Cancer
Keywords: Selumetinib; Tremelimumab; MEDI4736; Safety; Tolerability; Pharmacokinetics; Patients with advanced solid tumours; Disease progression
MeSH Terms: conditions — Lung Neoplasms; Melanoma; Breast Neoplasms; Colorectal Neoplasms; Biliary Tract Neoplasms; Disease Progression | interventions — AZD 6244; durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose escalation: Selumetinib+MEDI4736 (Experimental): An oral formulation of selumetinib will be administered in combination with an IV dose of MEDI4736. 4 cohorts of double combination (Selumetinib+MEDI4736).
  The decision to escalate to the next dose level/cohort will be made by the Safety Review Committee (SRC) following the completion of the dose limiting toxicity (DLT) assessment period for at least 3 evaluable patients in each cohort.
  Interventions: Drug: Selumetinib; Drug: MEDI4736
- Mandatory paired biopsy expansion cohort: Selumetinib+MEDI4736 (Experimental): One or more independent mandatory paired biopsy expansion cohorts for double combination treatment will start after safety and tolerability have been established for the relevant dose. It will be tumour-type specific for double combination, the tumor type will be determined from emerging data.
  Interventions: Drug: Selumetinib; Drug: MEDI4736
- Dose escalation: Selumetinib+MEDI4736+tremelimumab (Experimental): An oral formulation of selumetinib will be administered in combination with an IV dose of MEDI4736 and an IV dose of tremelimumab.
  For triple combination treatment, the starting dose of selumetinib (DL1) will be determined by the SRC based on emerging data from dose escalation cohorts of double combination treatment.
  Interventions: Drug: Selumetinib; Drug: MEDI4736; Drug: Tremelimumab
- Mandatory paired biopsy expansion cohort: triple combination (Experimental): One or more independent mandatory paired biopsy expansion cohorts for triple combination treatment will start after safety and tolerability have been established for the relevant dose. It will be tumour-type specific for triple combination, the tumor type will be determined from emerging data.
  Interventions: Drug: Selumetinib; Drug: MEDI4736; Drug: Tremelimumab

INTERVENTIONS:
Drug: Selumetinib — Selumetinib oral
Drug: MEDI4736 — MEDI4736 IV
Drug: Tremelimumab — Tremelimumab, IV
  Arms: Dose escalation: Selumetinib+MEDI4736+tremelimumab; Mandatory paired biopsy expansion cohort: triple combination

SUMMARY:
This is a Phase I, open-label, multi-centre, drug combination study of double and triple combination oral selumetinib (AZD6244 Hyd-sulfate) plus intravenous (IV) MEDI4736 and oral selumetinib plus IV MEDI4736 and IV tremelimumab in patients with advanced solid tumours.

DETAILED DESCRIPTION:
This is a Phase I, open-label, multi-centre, drug combination study of double and triple combination oral selumetinib (AZD6244 Hyd-sulfate) plus intravenous (IV) MEDI4736 and oral selumetinib plus IV MEDI4736 and IV tremelimumab in patients with advanced solid tumours refractory to standard therapy or for which no standard therapy exists. The safety, tolerability, and preliminary anti-tumour activity of ascending doses of Selumetinib (AZD6244 Hyd-sulfate) in Combination with MEDI4736 and Selumetinib in Combination with MEDI4736 and Tremelimumab will be investigated. Once safety and tolerability have been established for the relevant dose, expansion cohorts will commence in order to further evaluate safety, tolerability, and provide a preliminary evaluation of the mechanism of action and anti-tumour activity of the drug combination. Mandatory paired biopsy expansion cohorts will be tumour-type specific. Expansion cohorts will open independently for double and triple combination treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (eg, Health Insurance Portability and Accountability Act in the US, EU Data Privacy Directive in the EU) obtained from the patient prior to performing any protocol-related procedures, including pre-screening and screening evaluations
2. Age ≥18 years at time of study entry
3. Histological or cytological confirmation of locally advanced (stage IIIB) or metastatic (stage IV) solid tumours refractory to standard therapy or for which no standard therapy exists
4. World Health Organisation Eastern Cooperative Oncology Group (ECOG) performance status 0-1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks
5. At least 1 lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated assessment as per Response Evaluation Criteria in Solid Tumours (RECIST criteria v1.1)
6. Female patients and males with partners of childbearing potential should be using highly effective contraceptive measures. Females should not be breastfeeding and must have a negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential by fulfilling 1 of the criteria below at screening.

   * Postmenopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women <50 years old would be considered postmenopausal if they have been amenorrheic for the past 12 months or more following cessation of exogenous hormonal treatments. The levels of luteinising hormone (LH) and follicle stimulating hormone (FSH) must also be in the postmenopausal range (as per the institution)
   * Documentation of irreversible surgical sterilisation by hysterectomy and / or bilateral oophorectomy and/or bilateral salpingectomy but not tubal ligation
7. Male patients should be willing to use barrier contraception ie, condoms plus spermicide
8. Mandatory provision of tumour tissue sample available at study entry for exploratory biomarker research. Cytology samples for this exploratory biomarker research will not be acceptable
9. Patients must have mCRC and, if MSI status is known, non-high MSI status. MSI status will be evaluated based on previous results of local MSI testing, if available. Patients with known MSI-high status will be excluded; patients with MSS, MSI-low, or unknown MSI status may be enrolled

Exclusion Criteria:

Patients must not enter the study if any of the following exclusion criteria are fulfilled

1. Previous enrolment in the present study
2. Treatment with any of the following:

   * Cytotoxic chemotherapy or other anticancer drugs within 28 days of the 1st dose of study treatment or any investigational agents within 5 half-lives of the product
   * MEDI4736 or selumetinib in the present study (ie, dosing with MEDI4736 or selumetinib previously initiated in this study)
   * Major surgical procedure, (excluding placement of vascular access) or significant traumatic injury within 4 weeks of the 1st dose of study treatment, or have an anticipated need for major surgery during the study
   * Palliative radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the 1st dose of study treatment
   * Prior exposure to immune-mediated therapy, including, but not limited to, other anti-CTLA- 4 (Cytotoxic T-lymphocyte antigen-4), anti-PD-1 (Programmed cell death 1), anti-PD-L1 (Programmed cell death ligand 1), or anti-PD-L2 (Programmed cell death ligand 2) antibodies, including therapeutic anticancer vaccines
   * Receipt of live attenuated vaccine within 30 days prior to the first dose of IP
   * Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
3. Any unresolved toxicity NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis and may be included after consultation with the medical monitor
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with selumetinib, MEDI4736 or tremelimumab may be included after consultation with the medical monitor
4. History of leptomeningeal carcinomatosis and brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have a CT / MRI of the brain prior to study entry
5. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], celiac disease, irritable bowel disease, or other serious GI (Gastrointestinal) chronic conditions associated with diarrhoea, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [eg, granulomatosis with polyangiitis, Graves' disease; rheumatoid arthritis, hypophysitis, uveitis]) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment
6. History of active primary immunodeficiency
7. Current or prior use of immunosuppressive medication within 14 days before the 1st dose of MEDI4736. The following are exceptions to this criterion:

   * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection)
   * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
   * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
8. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, renal transplant, active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol or active infection including hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) or known history of clinical diagnosis of tuberculosis
9. Screening for chronic conditions is not required
10. Any of the following cardiac criteria:

    * Any factors that increase the risk of QT(ECG interval measured from the onset of the QRS complex to the end of the T wave) interval corrected for heart rate (QTc) prolongation or risk of arrhythmic events (eg, heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age) or mean QTc >470 msec
    * Uncontrolled hypertension (eg, BP ≥150/95 mmHg despite medical therapy)
    * Acute coronary syndrome within 6 months prior to starting treatment
    * Angina Canadian Cardiovascular Society Grade II-IV (despite medical therapy)
    * Symptomatic heart failure (New York Heart Association II-IV)
    * Prior or current cardiomyopathy
    * Baseline LVEF (Left ventricular ejection fraction) <55% measured by echocardiography or MUGA. Appropriate correction to be used if a MUGA is performed.
    * Atrial fibrillation with a ventricular rate >100 beats per minute at rest
    * Severe valvular heart disease
11. Any of the following ophthalmic criteria:

    * Current or past history of central serous retinopathy, detachment of retinal pigmented epithelium, or retinal vein occlusion
    * Intraocular pressure (IOP) >21 mmHg
    * Uncontrolled glaucoma (irrespective of IOP)
12. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

    * Absolute neutrophil count <1.5 x 109/L
    * Platelet count <100 x 109/L
    * Haemoglobin <90 g/L
    * Alanine aminotransferase >2.5 x ULN (upper limit of normal) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
    * Aspartate aminotransferase >2.5 x ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
    * Serum bilirubin ≤1.5 x ULN. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinaemia [predominantly unconjugated bilirubin] in the absence of evidence of haemolysis or hepatic pathology), who will be allowed in consultation with their physician
    * Creatinine clearance <50 mL/min (calculated by Cockcroft and Gault equation). Confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN
13. Refractory nausea and vomiting, chronic GI diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of selumetinib
14. History of hypersensitivity to active or inactive excipients of MEDI4736 or selumetinib or drugs with a similar chemical structure or class to MEDI4736 or selumetinib
15. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements
16. Involvement in the planning and conduct of the study (applies to both AZ staff or staff at the study site)
17. Previous allogeneic bone marrow transplant
18. Body weight <30 kg

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of Adverse Events | From screening until approximately 30 days after last dose of study drug at disease progression
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of safety laboratory tests | From screening until approximately 30 days after last dose of study drug at disease progression
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of blood pressure (BP) | From screening until approximately 30 days after last dose of study drug at disease progression
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of Electrocardiogram (ECG) | From screening until approximately 30 days after last dose of study drug at disease progression
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of physical examinations | From screening until approximately 30 days after last dose of study drug at disease progression
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of Echocardiogram (ECHO) | From screening until approximately 30 days after last dose of study drug at disease progression
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of pulse | From screening until approximately 30 days after last dose of study drug at disease progression
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of body temperature | From screening until approximately 30 days after last dose of study drug at disease progression
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of respiratory rate | From screening until approximately 30 days after last dose of study drug at disease progression
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of Multigated Acquisition (MUGA) | From screening until approximately 30 days after last dose of study drug at disease progression
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of Ophthalmic examination (best corrected visual acuity) | From screening until approximately 30 days after last dose of study drug at disease progression
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of Ophthalmic examination (Intraocular pressure) | From screening until approximately 30 days after last dose of study drug at disease progression
Safety and tolerability of Selumetinib in combination with MEDI4736, and in combination with MEDI4736+ tremelimumab by assessment of Ophthalmic examination (slit lamp fundoscopy) | From screening until approximately 30 days after last dose of study drug at disease progression

SECONDARY OUTCOMES:
Long-term tolerated dose and exposure predicted to result in biological activity (including but not limited to Response Evaluation Criteria in Solid Tumours (RECIST) | From screening until 30 days after last dose of study drug at disease progression, approximately 6 months however there is no maximum duration of treatment
Objective response rate (ORR) | From screening until 30 days after last dose of study drug at disease progression, approximately 6 months however there is no maximum duration of treatment
Change in tumour size | From screening until 30 days after last dose of study drug at disease progression, approximately 6 months however there is no maximum duration of treatment
Best Objective Response (BoR) | From screening until 30 days after last dose of study drug at disease progression, approximately 6 months however there is no maximum duration of treatment
Duration of Response (DoR) | From screening until 30 days after last dose of study drug at disease progression, approximately 6 months however there is no maximum duration of treatment
Progression-free survival (PFS) | From screening until 30 days after last dose of study drug at disease progression, approximately 6 months however there is no maximum duration of treatment
Overall survival (OS) | From screening until 30 days after last dose of study drug at disease progression, approximately 6 months however there is no maximum duration of treatment
MEDI4736 and/or tremelimumab anti-drug antibody (ADA) level in Plasma | From screening until 30 days after last dose of study drug at disease progression, approximately 6 months however there is no maximum duration of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pasi A. Jänne, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Las Vegas, Nevada
  - Research Site, New Brunswick, New Jersey
  - Research Site, Charlotte, North Carolina
  - Research Site, Pittsburgh, Pennsylvania